CLINICAL TRIAL: NCT05024344
Title: Erector Spinae Plane Block Versus Control for Pain Control Following Percutaneous Nephrolithotomy: A Randomized, Double-Blind, Placebo Controlled Study
Brief Title: ESP Block vs Control for Pain Control Following Percutaneous Nephrolithotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ANES-01-072021
Record Dates: First submitted 2021-08-02; First posted 2021-08-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Nephrolithotomy, Percutaneous
MeSH Terms: interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ESP Group (Active Comparator): One 30mL syringe containing 30mL of 0.5% ropivacaine and 4 mg of dexamethosone-
  Interventions: Procedure: Erector Spinae Plane Block; Drug: Ropivacaine 0.5% Injectable Solution; Drug: Dexamethasone
- Sham Group (Sham Comparator): One 30mL syringe containing 30mL of preservative free normal saline
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The Anesthesiologist will use ultrasound-guided technique and inject 30mL of 0.5% ropivacaine with 4 mg of dexamethasone or saline placebo control into the erector spinae muscle, superficial to the tips of the thoracic transverse processes
Drug: Ropivacaine 0.5% Injectable Solution — The Anesthesiologist will use ultrasound-guided technique and inject 30mL of 0.5% ropivacaine with 4 mg of dexamethasone or saline placebo control into the erector spinae muscle, superficial to the tips of the thoracic transverse processes
  Arms: ESP Group
Drug: Dexamethasone — The Anesthesiologist will use ultrasound-guided technique and inject 30mL of 0.5% ropivacaine with 4 mg of dexamethasone or saline placebo control into the erector spinae muscle, superficial to the tips of the thoracic transverse processes
  Arms: ESP Group

SUMMARY:
The purpose of this study is to investigate the use of the erector spinae (ESP) block in reducing the morphine milligram equivalent (MME) consumption post percutaneous nephrolithotomy. Objectives:

1. - Determine if there is a significant effect on post percutaneous nephrolithotomy MME consumption with the usage of an ESP block vs. saline control.
2. - Determine if there is a significant effect on reported pain levels with the use of an ESP block vs. saline control in post percutaneous nephrolithotomies.

DETAILED DESCRIPTION:
This is a double-blind, randomized control trial involving 128 subjects undergoing an elective percutaneous nephrolithotomy. All subjects who meet all inclusion and exclusion criteria will be equally randomized on the day of the procedure by operating room pharmacy into either the ESP block or the control block. An interim analysis at the sample size required for a large effect size (n = 52, with n = 26 in each treatment arm) will be performed. In order to blind the anesthesiologist performing the block, the control arm will be equally randomized by the pharmacist at the time of distributing the pre-filled syringes for the ESP block procedure. Randomization will occur with the use of a random number generator with 1:1 ESP:Control allocation ratio.

Subjects will be followed at Pre-op and the 24-h, 48-h, 7 days and 30 days post operatively to assess the quality of recovery utilizing the Quality of Recovery-15 (QoR-15) questionnaire, VAS pain scale, and opioid consumption. Intraoperative MMEs, PACU MMEs, total MME's, FLACC scores at 30 minutes/1 hour VAS scores at 1 hour/2 hours/6 hours/24 hours, PACU LOS, hospital LOS, time to first flatus will be documented in patient chart, reviewed by study personnel and uploaded into a password protected database on the UTMCK server.

All aspects of the study and consent forms will be IRB approved prior to implementation. Potential candidates will be selected for consent based on chart review and surgery scheduling.

* The Surgeon will initially approach potential subjects and provide them with a copy of the consent form to take home and read prior to pre-anesthesia testing.
* At the subject's pre-anesthesia testing appointment, the research staff will explain the risks and benefits of the study, answer any questions, and obtain consent to participate.
* The Biostatistician will randomize the subjects with a random number generator. Once randomized, a blinded package labeled "ESP" or "Control" will be delivered to the regional anesthesia team containing the following:

ESP

Active group:

1. One 30mL syringe containing 29mL of 0.5% ropivacaine and 4mg of dexamethasone- labeled "ESP Block"
2. One 30mL syringe containing 30mL of preservative free normal saline- labeled "wound infiltration" Sham group

1. One 30mL syringe containing 30mL of 0.5% ropivacaine- labeled "wound infiltration" 2. One 30mL syringe containing 30mL of preservative free normal saline- labeled "ESP Block"

* The pharmacist will create a table pre-populated with the randomization assignments with space to fill out patient information and medication information on the day of surgery. This chart will be in paper form and kept in a research binder in the OR pharmacy. When a patient is consented for the RCT, the treatment group will be chosen based on the numbers assigned a priori. Each qualifying patient will be documented on the subsequent row in the table, maintaining the original order of randomization as dictated by the statistician. Based on the assignment, the pharmacy technician will be instructed as to which products to make in the sterile hood. The pharmacist will verify that the products were made appropriately and will label the syringes according to assignment.
* Operating room pharmacy will hand the anesthesiologist a blinded package with one prefilled syringe for the regional block that will either contain 30mL of 0.5% ropivacaine with 4mg of dexamethasone or preservative free normal saline.
* The regional anesthesiologist will perform the ESP block using standard protocols and procedures.
* Age, BMI, duration of operation, EBL, intraoperative MMEs, PACU MMEs, 48 hours post-operative MMEs, total MME's, FLACC scores at 30 minutes/1 hour VAS scores at 1 hour/2 hours/6 hours/24 hours, PACU LOS, hospital LOS, time to first flatus will be documented in patient chart and reviewed by study personnel.
* QoR-15, MME consumption, and VAS will be assessed at Pre-op, 24-h, 48-h, 7 and 30 days by study staff. Data will be uploaded into a database kept on secured password protected computers on the UTMCK server.
* All patient identifiers will be removed prior to data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male and female greater than or equal to 18 years of age and undergoing non-emergent percutaneous nephrolithotomy Monday through Friday between the hours of 6:00AM and 4:00PM.
* Female participants of childbearing potential will be required to provide a negative pregnancy test.
* Ability to understand and teach back consent for the procedure.
* Willingness to sign consent for procedure.
* English speaking.

Exclusion Criteria:

* Emergent surgery status.
* Local infection
* Allergy to local anesthetics.
* Recreational drug use.
* Inability to provide informed consent.
* Pregnancy or breastfeeding.
* History of Guillain-Barre' Syndrome.
* Underlying medical conditions that would post a significant risk to the patient.
* Opioid use >90 days in the year leading up to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption (MME) | First 24 hours postoperative
  Opioid consumption (MME) in the first 24 hours postoperative

SECONDARY OUTCOMES:
Hospital LOS | Number of days in hospital (inpatient) from day of surgery (day 1) until discharge post-surgery in 24 hour increments up to 30 days
  Hospital length of stay
VAS score | First 24 hours after surgery.
  Mean Visual Analog Scale (VAS) score in the first 24 hours after surgery. VAS measures the amount of pain that a patient feels ranging across a continuum from none(0) to an extreme amount of pain(10) on a chart.
Opioid use during first 24 hours after surgery | 24 hours
  MMEs (morphine milligram equivalent) administered during first 24 hours post surgery
QoR-15 | 24 hours, 48 hours, 7 days, and 30 days after surgery
  Quality of Recovery -15 at 24 hours, 48 hours, 7 days, and 30 days after surgery. QoR-15 measures how a patient feels they are recovering after surgery using a 15 item survey rated 0 (none of the time-poor) to 10 (all of the time-excellent).
Opioid use during 30 days post hospital discharge | 30 days
  MMEs administered/consumed during 30 day period post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jason Buehler, MD, Principal Investigator — University of Tennessee Medical Center
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dundar G, Gokcen K, Gokce G, Gultekin EY. The Effect of Local Anesthetic Agent Infiltration Around Nephrostomy Tract On Postoperative Pain Control After Percutaneous Nephrolithotomy: A single-centre, randomised, double-blind, placebocontrolled clinical trial. Urol J. 2018 Nov 17;15(6):306-312. doi: 10.22037/uj.v0i0.4145. PMID 29681047
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Tulgar S, Selvi O, Ozer Z. Clinical experience of ultrasound-guided single and bi-level erector spinae plane block for postoperative analgesia in patients undergoing thoracotomy. J Clin Anesth. 2018 Nov;50:22-23. doi: 10.1016/j.jclinane.2018.06.034. Epub 2018 Jun 23. No abstract available. PMID 29940470
- [Background] Kwon WJ, Bang SU, Sun WY. Erector Spinae Plane Block for Effective Analgesia after Total Mastectomy with Sentinel or Axillary Lymph Node Dissection: a Report of Three Cases. J Korean Med Sci. 2018 Nov 5;33(45):e291. doi: 10.3346/jkms.2018.33.e291. No abstract available. PMID 31044575
- [Background] Ibrahim M, Elnabtity AM. Analgesic efficacy of erector spinae plane block in percutaneous nephrolithotomy : A randomized controlled trial. Anaesthesist. 2019 Nov;68(11):755-761. doi: 10.1007/s00101-019-00673-w. Epub 2019 Oct 16. PMID 31620856
- [Background] Govender S, Mohr D, Van Schoor AN, Bosenberg A. The extent of cranio-caudal spread within the erector spinae fascial plane space using computed tomography scanning in a neonatal cadaver. Paediatr Anaesth. 2020 Jun;30(6):667-670. doi: 10.1111/pan.13864. Epub 2020 Apr 22. PMID 32267041
- [Background] Ugras MY, Toprak HI, Gunen H, Yucel A, Gunes A. Instillation of skin, nephrostomy tract, and renal puncture site with ropivacaine decreases pain and improves ventilatory function after percutaneous nephrolithotomy. J Endourol. 2007 May;21(5):499-503. doi: 10.1089/end.2006.0335. PMID 17523902
- [Result] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05024344/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05024344/ICF_001.pdf